CLINICAL TRIAL: NCT05253872
Title: The MELAcare Study: a Randomized Controlled Trial of a New Method for Surveillance of Melanoma Patients
Brief Title: The MELAcare Study: A New Method for Surveillance of Melanoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Sara Molgaard Hansen, Principal investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Melacare v1.0
Record Dates: First submitted 2022-01-24; First posted 2022-02-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Cutaneous Melanoma
Keywords: cutaneous melanoma; follow-up; nurse-led follow-up; skin self-examination; survivorship
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention arm will receive follow-up conducted by melanoma nurses, where the patients will get tools to cope with the melanoma diagnosis and structured training in skin self-examination
  Interventions: Other: The MelaCare intervention
- Control group (No Intervention): Patients in the control arm will receive clinical follow-up according to the current standard of care for their clinical stage.

INTERVENTIONS:
Other: The MelaCare intervention — The primary principles applied will be:
  * Meta-cognitive strategies and normalization of emotions
  * Self efficacy related to SSE and knowledge on when to seek a doctor for clinical examination
  The intervention will include 4 components:
  * An educational booklet
  * Doctor consultation to ensure correct SSE skills and compliance to the protocol
  * 3-5 sessions with a experienced and specially trained melanoma nurse
  * Use of patients' answers from the Patient Reported Outcome 'Functional Assessment of Cancer Treatment - Melanoma' (FACT-M) at the nurse sessions to address current emotional and/or physical sequelae.
  Arms: Intervention group

SUMMARY:
The aim of this study is to evaluate a new method of follow-up for patients with low and intermediate risk (stages IA-IIA) melanoma. The investigators will compare different tools for patient support and education combined with clinician supported skin self-examination (SSE) to the current standard-of-care. The hypothesis is that meta-cognitive strategies and clinician supported SSE can lower fear of cancer recurrence (FCR) and promote effective SSE on a regular basis without compromising the detection of new primary melanomas and/or metastases.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand Danish language
* Willing and able to give written informed consent
* Surgical treatment of a clinical stage IA-IIA melanoma within 3 months of inclusion

Exclusion Criteria:

* Advanced melanoma, clinical stages IIB, IIC, III, or IV
* Patients with high risk of a new primary melanoma (dysplastic nevus syndrome, or family history of melanoma)
* History of melanoma skin cancer prior to the index diagnosis
* Previous cancer, excluding non-melanoma skin cancer
* Comorbidity that makes skin self-examination impossible (e.g. physical or mental disabilities, dementia or decreased cognitive function)
* non-detection of sentinel node in IB and IIA patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence | The primary outcome will be evaluated at approx. 6-8 months after randomization.
  The primary outcome is the score of the validated 4-item Concerns About Recurrence Questionnaire (CARQ-4). A higher score indicates a higher level of FCR. A score of 12 or above is considered clinically relevant fear of cancer recurrence.
Fear of cancer recurrence | The primary outcome will be evaluated at approx. 12 months follow-up
  The primary outcome is the score of the validated 4-item Concerns About Recurrence Questionnaire (CARQ-4). A higher score indicates a higher level of FCR. A score of 12 or above is considered clinically relevant fear of cancer recurrence.
Fear of cancer recurrence | The primary outcome will be evaluated at approx. 24 months follow-up
  The primary outcome is the score of the validated 4-item Concerns About Recurrence Questionnaire (CARQ-4). A higher score indicates a higher level of FCR. A score of 12 or above is considered clinically relevant fear of cancer recurrence.

SECONDARY OUTCOMES:
Evaluation of change from baseline in depression score by the validated Patient Health Questionnaire-9 (PhQ-9) | Depression score will be evaluated at approx. 6-8 months after randomization.
  The PhQ-9 has a scale from 0-27, and a higher score is associated with increase in depression severity
Evaluation of change from baseline in depression score by the validated Patient Health Questionnaire-9 (PhQ-9) | Depression score will be evaluated at approx. 12 months follow-up
  The PhQ-9 has a scale from 0-27, and a higher score is associated with increase in depression severity
Evaluation of change from in depression score by the validated Patient Health Questionnaire-9 (PhQ-9) | Depression score will be evaluated at 24 months follow-up
  The PhQ-9 has a scale from 0-27, and a higher score is associated with increase in depression severity
Evaluation of change from baseline in anxiety score by the validated General Anxiety Disorder-7 questionnaire (GAD-7) | Anxiety score will be evaluated at approx. 6-8 months after randomization.
  The GAD-7 has a scale from 0-21, and a higher score is associated with increase in anxiety severity.
Evaluation of change from baseline in anxiety score by the validated General Anxiety Disorder-7 questionnaire (GAD-7) | Anxiety score will be evaluated at approx.12 months follow-up
  The GAD-7 has a scale from 0-21, and a higher score is associated with increase in anxiety severity.
Evaluation of change from baseline in anxiety score by the validated General Anxiety Disorder-7 questionnaire (GAD-7) | Anxiety score will be evaluated at approx. 24 months follow-up
  The GAD-7 has a scale from 0-21, and a higher score is associated with increase in anxiety severity.
Evaluation of change from baseline in distress score by the validated distress thermometer | Distress score will be evaluated at approx. 6-8 months after randomization.
  The distress thermometer has a scale from 0-10, and a higher score is associated with increase in distress severity
Evaluation of change from baseline in distress score by the validated distress thermometer | Distress score will be evaluated at approx.12 months follow-up
  The distress thermometer has a scale from 0-10, and a higher score is associated with increase in distress severity
Evaluation of change from baseline in distress score by the validated distress thermometer | Distress score will be evaluated at approx. 24 months follow-up
  The distress thermometer has a scale from 0-10, and a higher score is associated with increase in distress severity
Evaluation of change from baseline in activation score by the validated patient activation measure | Activation measure will be evaluated at approx. 6-8 months after randomization.
  The patient activation measure has a 100-point scale, and a higher score is associated with increase in activation level
Evaluation of change from baseline in activation score by the validated patient activation measure | Activation measure will be evaluated at approx.12 months follow-up
  The patient activation measure has a 100-point scale, and a higher score is associated with increase in activation level
Evaluation of change from baseline in activation score by the validated patient activation measure | Activation measure will be evaluated at approx. 24 months follow-up
  The patient activation measure has a 100-point scale, and a higher score is associated with increase in activation level
Evaluation of change from baseline in health status by the validated Euroqol 5 dimensions, 3 levels questionnaire (EQ-5D-3L) | Health status will be evaluated at approx. 6-8 months after randomization.
  The EQ-5D-3L has a 3-level scale, and a higher level is associated with decrease in health status
Evaluation of change from baseline in health status by the validated Euroqol 5 dimensions, 3 levels questionnaire (EQ-5D-3L) | Health status will be evaluated at approx.12 months follow-up
  The EQ-5D-3L has a 3-level scale, and a higher level is associated with decrease in health status
Evaluation of change from baseline in health status by the validated Euroqol 5 dimensions, 3 levels questionnaire (EQ-5D-3L) | Health status will be evaluated at approx. 24 months follow-up
  The EQ-5D-3L has a 3-level scale, and a higher level is associated with decrease in health status
Evaluation of change from baseline in work ability by the validated work ability index | Work ability will be evaluated at approx. 6-8 months after randomization.
  The work ability index has a scale from 7-49, where higher scores indicates better work ability.
Evaluation of change from baseline in work ability by the validated work ability index | Work ability will be evaluated at approx.12 months follow-up
  The work ability index has a scale from 7-49, where higher scores indicates better work ability.
Evaluation of change from baseline in work ability by the validated work ability index | Work ability will be evaluated at approx. 24 months follow-up
  The work ability index has a scale from 7-49, where higher scores indicates better work ability.
Evaluation of the time and costs spend by the patients getting to and from the follow-up visits | Time and costs spend will be evaluated at approx. 6-8 months after randomization.
  The patients will fill in a study specific questionnaire informing time and money spent for transportation to and from the follow-up visits
Evaluation of the time and costs spend by the patients getting to and from the follow-up visits | Time and costs spend will be evaluated at approx.12 months follow-up
  The patients will fill in a study specific questionnaire informing time and money spent for transportation to and from the follow-up visits
Evaluation of the time and costs spend by the patients getting to and from the follow-up visits | Time and costs spend will be evaluated at approx. 24 months follow-up
  The patients will fill in a study specific questionnaire informing time and money spent for transportation to and from the follow-up visits
Evaluation of the number of extra clinical consultations with a doctor at the outpatient clinic | the number of extra clinical consultations with a doctor will be evaluated at approx. 6-8 months after randomization.
  The investigators will evaluate number of extra clinical consultations with a doctor the patients will attend at the outpatient clinic. The data will be collected using electronic patient journal.
Evaluation of the number of extra clinical consultations with a doctor at the outpatient clinic | the number of extra clinical consultations with a doctor will be evaluated at approx. 12 months follow-up
  The investigators will evaluate number of extra clinical consultations with a doctor the patients will attend at the outpatient clinic. The data will be collected using electronic patient journal.
Evaluation of the number of extra clinical consultations with a doctor at the outpatient clinic | the number of extra clinical consultations with a doctor will be evaluated at approx. 24 months follow-up
  The investigators will evaluate number of extra clinical consultations with a doctor the patients will attend at the outpatient clinic. The data will be collected using electronic patient journal.
Evaluation of the number of extra clinical consultations with a doctor at the outpatient clinic | the number of extra clinical consultations with a doctor will be evaluated at approx. 60 months follow-up
  The investigators will evaluate number of extra clinical consultations with a doctor the patients will attend at the outpatient clinic. The data will be collected using electronic patient journal.
Evaluation of the number and characteristics of new primary melanomas and/or recurrences | Number and characteristics of new primary melanoma and/or recurrences will be evaluated at approx. 6-8 months after randomization.
  The investigator will register any new melanomas and recurrences detected, and deaths. The data will be collected using medical records.
Evaluation of the number and characteristics of new primary melanomas and/or recurrences | Number and characteristics of new primary melanoma and/or recurrences will be evaluated at approx.12 months follow-up
  The investigator will register any new melanomas and recurrences detected, and deaths. The data will be collected using medical records.
Evaluation of the number and characteristics of new primary melanomas and/or recurrences | Number and characteristics of new primary melanoma and/or recurrences will be evaluated at approx. 24 months follow-up
  The investigators will register any new melanomas and recurrences detected, and deaths. The data will be collected using medical records.
Evaluation of the number and characteristics of new primary melanomas and/or recurrences | Number and characteristics of new primary melanoma and/or recurrences will be evaluated at approx. 60 months follow-up
  The investigators will register any new melanomas and recurrences detected, and deaths. The data will be collected using medical records.
Evaluation of time to diagnosis of a new primary melanoma and/or recurrence | Time to diagnosis of a new primary melanoma and/or recurrence will be evaluated at approx. 6-8 months after randomization.
  The investigators will evaluate time to diagnosis of a new melanomas using Breslows thickness as a proxy for time, and time to diagnosis recurrence measured by type of recurrence (local, regional or distant). The data will be collected using medical records.
Evaluation of time to diagnosis of a new primary melanoma and/or recurrence | Time to diagnosis of a new primary melanoma and/or recurrence will be evaluated at approx. 12 months follow-up
  The investigators will evaluate time to diagnosis of a new melanomas using Breslows thickness as a proxy for time, and time to diagnosis recurrence measured by type of recurrence (local, regional or distant). The data will be collected using medical records.
Evaluation of time to diagnosis of a new primary melanoma and/or recurrence | Time to diagnosis of a new primary melanoma and/or recurrence will be evaluated at approx. 24 months follow-up
  The investigators will evaluate time to diagnosis of a new melanomas using Breslows thickness as a proxy for time, and time to diagnosis recurrence measured by type of recurrence (local, regional or distant). The data will be collected using medical records.
Evaluation of time to diagnosis of a new primary melanoma and/or recurrence | Time to diagnosis of a new primary melanoma and/or recurrence will be evaluated at approx. 60 months follow-up
  The investigators will evaluate time to diagnosis of a new melanomas using Breslows thickness as a proxy for time, and time to diagnosis recurrence measured by type of recurrence (local, regional or distant). The data will be collected using medical records.
Evaluation of health care costs of the new follow-up program compared to the current | Health care costs evaluation will be evaluated at approx. 60 months follow-up
  We will evaluate the health care cost of new follow-up program compared to the current. Data will be collected using national registries.
Evaluation of the number of extra scans: Magnetic Resonance Imaging (MRI), computed tomography (CT), ultrasound, or positron emission tomography/computed tomography (PET/CT) | the number of extra scans will be evaluated at approx. 6-8 months after randomization.
  The investigators will evaluate number of extra scans. The data will be collected using electronic patient journal.
Evaluation of the number of extra scans: Magnetic Resonance Imaging (MRI), computed tomography (CT), ultrasound, or positron emission tomography/computed tomography (PET/CT) | the number of extra scans will be evaluated at approx. 12 months follow-up
  The investigators will evaluate number of extra scans. The data will be collected using electronic patient journal.
Evaluation of the number of extra scans: Magnetic Resonance Imaging (MRI), computed tomography (CT), ultrasound, or positron emission tomography/computed tomography (PET/CT) | the number of extra scans will be evaluated at approx. 24 months follow-up
  The investigators will evaluate number of extra scans. The data will be collected using electronic patient journal.
Evaluation of the number of extra scans: Magnetic Resonance Imaging (MRI), computed tomography (CT), ultrasound, or positron emission tomography/computed tomography (PET/CT) | the number of extra scans will be evaluated at approx. 60 months follow-up
  The investigators will evaluate number of extra scans. The data will be collected using electronic patient journal.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet R Hölmich, Professor, Study Chair — Herlev and Gentofte Hospital
Locations (1):
- Herlev and Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
There are no plan to share IPD with other researchers.

REFERENCES:
- [Derived] Hansen SM, Johansen C, Kasparian NA, Grand MK, Bidstrup PE, Holmich LR. Employing skin self-examination and fear of cancer recurrence management in early-stage melanoma follow-up: evaluation of the MELACARE intervention in a randomised controlled trial. J Cancer Surviv. 2025 Jun 12. doi: 10.1007/s11764-025-01841-1. Online ahead of print. PMID 40504479